CLINICAL TRIAL: NCT01532843
Title: Lowering Viral Load With Nucleos(T)Ide Analogues Prior to Peginterferon Alfa-2b Treatment to Increase Sustained Response in HBeAg-positive Chronic Hepatitis B (PEGON-study)
Brief Title: Lowering Viral Load With Nucleos(T)Ide Analogues Prior to Peginterferon Treatment to Ncrease Sustained Response in CHB
Acronym: PEGON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBV 11-02
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; sustained response; peginterferon; nucleos(t)ide analogues
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PegIFN alfa-2b + nucleos(t)ide analogue (Active Comparator): Peginterferon alfa-2b 1.5 μg/kg per week s.c. for 48 weeks in addition to standard nucleos(t)ide analogue treatment
  Interventions: Drug: PegIFN alfa-2b
- Nucleos(t)ide analogue (No Intervention): Continuation of Nucleos(t)ide analogue mono-therapy

INTERVENTIONS:
Drug: PegIFN alfa-2b — Peginterferon alpha-2b 1.5 μg/kg per week s.c.for 48 weeks
  Other Names: Pegintron
  Arms: PegIFN alfa-2b + nucleos(t)ide analogue

SUMMARY:
Treatment with a nucleoside analogue and subsequent viral decline has shown to partially restore immune hyporesponsiveness in chronic hepatitis B patients. Recent pilot studies investigating whether the effect of lowering viral load with nucleoside analogue therapy prior to the initiation of peginterferon results in higher sustained off-treatment responses showed contradictory findings.

The aim of this study is to investigate sustained off-treatment response to peginterferon alfa-2b in chronic HBeAg-positive hepatitis B patients who are pretreated with nucleos(t)ide analogues, thereby lowering viral load

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (HBsAg positive > 6 months)
* HBeAg positive, anti-HBe negative within 4 weeks prior to initiation of peginterferon alfa-2b
* HBV DNA < 2000 IU/ml within one month prior to initiation of peginterferon alfa-2b after a minimum of 12 months treatment with either Entecavir (one of all 3 brands) or Tenofovir
* ALT < 5x ULN
* Compensated liver disease
* Age ≥ 18 years and ≤ 70 years
* Written informed consent

Exclusion Criteria:

* Treatment with any investigational drug within 30 days of entry to this protocol
* Treatment with Telbivudine
* Severe hepatitis activity as documented by ALT > 5 x ULN
* History of decompensated cirrhosis (defined as jaundice in the presence of cirrhosis, ascites, bleeding gastric or esophageal varices or encephalopathy)
* Pre-existent neutropenia (neutrophils < 1,500/mm3) or thrombocytopenia (platelets < 90,000/mm3)
* Co-infection with hepatitis C virus or human immunodeficiency virus (HIV)
* Other acquired or inherited causes of liver disease: alcoholic liver disease, obesity induced liver disease, drug related liver disease, auto-immune hepatitis, hemochromatosis, Wilson's disease or alpha-1 antitrypsin deficiency
* Alpha fetoprotein > 50 ng/ml
* Hyper- or hypothyroidism (subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met)
* Immune suppressive treatment within the previous 6 months
* Contra-indications for alfa-interferon therapy like suspected hypersensitivity to interferon or Peginterferon or any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study.
* Pregnancy, breast-feeding
* Other significant medical illness that might interfere with this study: significant pulmonary dysfunction in the previous 6 months, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g. HIV positivity, auto-immune diseases, organ transplants other than cornea and hair transplant)
* Any medical condition requiring, or likely to require chronic systemic administration of steroids, during the course of the study
* Substance abuse, such as alcohol (> 80 g/day), I.V. drugs and inhaled drugs in the past 2 years.
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sustained response | at week 72
  Sustained response to therapy, defined as the combined presence of HBeAg seroconversion and HBV DNA < 200 IU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD PHD, Principal Investigator — Erasmus MC, University Medical Center Rotterdam
Locations (4):
- China (3):
  - Ruijin Hospital "Jiaolong University", Shanghai
  - Public Health Center "Fu Dan University", Shanghai
  - Zhong Shan Hospital "Fu Dan University", Shanghai
- Erasmus MC, University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brakenhoff SM, de Knegt RJ, Oliveira J, van der Eijk AA, van Vuuren AJ, Hansen BE, Janssen HLA, de Man RA, Boonstra A, Sonneveld MJ. Levels of Antibodies to Hepatitis B Core Antigen Are Associated With Liver Inflammation and Response to Peginterferon in Patients With Chronic Hepatitis B. J Infect Dis. 2022 Dec 28;227(1):113-122. doi: 10.1093/infdis/jiac210. PMID 35599306
- [Derived] Liem KS, van Campenhout MJH, Xie Q, Brouwer WP, Chi H, Qi X, Chen L, Tabak F, Hansen BE, Janssen HLA. Low hepatitis B surface antigen and HBV DNA levels predict response to the addition of pegylated interferon to entecavir in hepatitis B e antigen positive chronic hepatitis B. Aliment Pharmacol Ther. 2019 Feb;49(4):448-456. doi: 10.1111/apt.15098. PMID 30689258
- [Derived] Chi H, Hansen BE, Guo S, Zhang NP, Qi X, Chen L, Guo Q, Arends P, Wang JY, Verhey E, de Knegt RJ, Xie Q, Janssen HLA. Pegylated Interferon Alfa-2b Add-on Treatment in Hepatitis B Virus Envelope Antigen-Positive Chronic Hepatitis B Patients Treated with Nucleos(t)ide Analogue: A Randomized, Controlled Trial (PEGON). J Infect Dis. 2017 Apr 1;215(7):1085-1093. doi: 10.1093/infdis/jix024. PMID 28329061